CLINICAL TRIAL: NCT02524119
Title: A Phase Ib/II Study of LEE011 and Chemoembolization In Patients With Advanced Hepatocellular Carcinoma
Brief Title: LEE001 and Chemoembolization In Patients With Advanced Hepatocellular Carcinoma
Acronym: LEE001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: This study was terminated after the sponsor withdrew our support
Sponsor: University of Texas Southwestern Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Muhammad Beg, Associate Professor of Medicine, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 052015-073
Record Dates: First submitted 2015-07-30; First posted 2015-08-14 (Estimated); Results first posted 2021-02-01 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — ribociclib; Chemoembolization, Therapeutic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- LEE001 with Chemoembolization (Experimental): A total of 40 patients will be enrolled and undergo chemoembolization. Patients will receive LEE011 (600 mg PO once daily, 3 weeks on/1 week off) on Day 1 with chemoembolization. Patients can receive a total of 4 chemoembolization treatments within 6 month following first treatment as needed to treat initial HCC lesion.
  Interventions: Drug: LEE011; Procedure: Chemoembolization

INTERVENTIONS:
Drug: LEE011 — 600 mg PO once daily will be given orally on days 1-21 of a 28 day cycle (3 weeks on / 1 week off) :until disease progression, unacceptable toxicity, death, or discontinuation from the study treatment due to any other reason
Procedure: Chemoembolization — Patients will be treated with chemoembolization once every 4 weeks with up to 4 total chemoembolizations within the first 6 months from the initial chemoembolization.

SUMMARY:
The purpose of this study is determine whether the combination therapy with LEE011 and chemoembolization in patients with locally advanced Hepatocellular Carcinoma not amenable to curative therapies will provide greater efficacy than chemoembolization alone with a tolerable safety profile.

DETAILED DESCRIPTION:
Single-arm, single-institution, non-randomized, open-label phase II study to determine the efficacy and safety of treatment with LEE011 and chemoembolization in patients with advanced HCC (Hepatocellular Carcinoma) not amenable to curative therapies. A total of 40 patients will be enrolled and undergo chemoembolization. Patients will receive LEE011 (600 mg PO once daily, 3 weeks on/1 week off) on Day 1 with chemoembolization. Patients can receive a total of 4 chemoembolization treatments within 6 month following first treatment as needed to treat initial HCC (Hepatocellular Carcinoma) lesion.

Progression free survival will be based on tumor assessment using RECIST 1.1 criteria (Response Evaluation Criteria in Solid Tumors) Patients will receive trial treatment until disease progression, unacceptable toxicity, death or discontinuation from the study treatment for any other reason. Patients will be followed for survival regardless of treatment discontinuation for any reason.

The study will include men and women with locally advanced HCC (Hepatocellular Carcinoma) not amenable to curative therapy who have received no prior therapy for advanced disease.

Investigational Therapy:

LEE011 oral (3 weeks on/1 week off) in combination with chemoembolization.

Efficacy Assessments:

1. Dynamic contrasted abdominal computed tomography or magnetic resonance imaging will be done at baseline, every 8 weeks, and every 3 months thereafter following initial chemoembolization.
2. Chest CT imaging as clinically indicated
3. Survival status every 12 months (or earlier if required) regardless of treatment discontinuation reason

Data Analysis:

The primary endpoint of the trial will be progression free survival (PFS) of HCC patients. PFS is defined to be the time from initiation of treatment to progression or death without evidence of progression. For cases without documentation of progression, follow-up will be censored at the date of last disease assessment without progression, unless death occurs within 4 months following the date of last progression-free, in which case death will be counted as an event. The historical median PFS for TACE (Transcatheter arterial chemoembolization) alone is 8-10 months. This study will target a hazard ratio of 0.69 with an 80% power and a one-sided significance level of 10%. Assuming a 24-month accrual and an 18-month follow-up period the study requires 38 patients initiating LEE011 treatment with the median PFS for TACE alone is 8 months, and 41 patients with the median PFS for TACE(Transcatheter arterial chemoembolization) alone is 10 months. PFS will be estimated using the Kaplan-Meier method, and Greenwood's formula will be used to calculate the standard error of the corresponding Kaplan-Meier estimate and 95% confidence interval. Survival curves will be estimated using Kaplan-Meier methodology.

Secondary endpoints of efficacy are to evaluate OS (Overall Survival). The statistical methods used for the analysis of PFS will be used for the analysis of OS.

Other secondary objectives will include description of toxicity of the therapy regimen. These data will be analyzed separately. The safety analyses will be performed on all patients who receive any dose of therapy. Adverse events will be described using the NCI CTCAE v 4.03 criteria (ctep.cancer.gov/forms.CTCAEv4.pdf). Frequency and severity of adverse events according to the NCI CTCAE ) v 4.03 (Common Terminology Criteria for Adverse Events) body system and severity criteria will be described. In addition, frequency of Grade 3 or 4 adverse events will be described separately. Causality will also be noted. Adverse events will be recorded for up to 1 year following discontinuation from study. Response rate and toxicity rate will be estimated using an exact binomial method along with the 95% confidence interval

ELIGIBILITY:
Inclusion Criteria:

1. Patient must have a histologically confirmed diagnosis of RB positive hepatocellular carcinoma
2. Patients must have HCC limited to the liver. There must be no clinical or radiographic evidence of extrahepatic HCC. Portal lymphadenopathy is permitted as lymphadenopathy is commonly associated with cirrhosis unrelated to malignancy;
3. Absence of occlusive main portal vein thrombus, branch venous thrombus is allowed;
4. Patients with locally advanced HCC not eligible for curative therapies;
5. Age ≥ 18 years;
6. Child-Pugh Score A or B7;
7. ECOG (Eastern Cooperative Oncology Group) Performance score of 0-2;
8. Life expectancy greater than 6 months;
9. Following baseline laboratory values:
10. Total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well-documented Gilbert's Syndrome;
11. INR (international normalized ratio) ≤ 1.7;
12. Hgb ≥ 9.0 g/dl;
13. Alkaline Phosphatase, AST (Aspartate Aminotransferase), ALT (Alanine Aminotransferase) <7 times ULN;
14. Platelet count ≥ 75,000/mm3;
15. Serum creatinine ≤ 1.5 mg/dL or creatinine clearance ≥ 50 mL/min;
16. Absolute neutrophil ≥ 1,500 cells/mm3;
17. Potassium, total calcium (corrected for serum albumin), magnesium, and phosphorus within normal limits for the institution or corrected to within normal limits with supplements before first dose of study medication
18. Sodium >130 meq/L;
19. Women of childbearing potential must have a negative pregnancy test;
20. Prior therapy is allowed provided the following are met: at least 4 weeks since prior locoregional therapy including surgical resection, chemoembolization, radiotherapy, or ablation. Provided target lesion has increased in size by 25% or more or the target lesion was not treated with locoregional therapy;
21. Must be able to swallow LEE011 capsules.

Exclusion Criteria:

1. Patient who received any CDK4/6 inhibitor (cyclin-dependent kinase 4);
2. Patient who has received previous systemic therapy;
3. Patients with central nervous system (CNS) involvement, unless they meet ALL of the following criteria:
4. At least 4 weeks from prior therapy completion (including ration and/or surgery) to starting the study treatment;
5. Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases;
6. Clinically significant, uncontrolled heart disease and/or recent events including any of the following:
7. History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) or symptomatic pericarditis within 12 months prior to screening;
8. History of documented congestive heart failure (New York Heart Association functional classification III-IV);
9. Documented cardiomyopathy;
10. Patient has a left ventricular ejection fraction <50% as determined by MUGA (Multi Gated Acquisition scan) or ECHO at screening;
11. History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrythmias, or conduction abnormality within 12 months of screening;
12. Bradycardia (heart rate <50 at rest), by ECG or pulse, at screening;
13. Congenital long QT syndrome or family history of long QT syndrome;
14. Systolic Blood Pressure (SBP) >160 or <90 mm Hg;
15. On screening inability to determine the QTcF (Fridericia Correction Formula) interval on the ECG (i.e.: Unreadable or Not Interpretable) or QTcF > 450 msec (using Fridericia's correction). All as determined by screening ECG (mean of triplicate ECGs);
16. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to treatment (see appendix 1 for details):
17. Known strong inducers or inhibitors of CYP3A4/5 (a member of the cytochrome P450), including grapefruit, grapefruit hybrids, pomelo, star-fruit, and Seville oranges;
18. That have a known risk to prolong the QT interval or induce Torsades de Pointes
19. Herbal preparations/medications, dietary supplements;
20. That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5;
21. Tumor involvement > 50% of the liver;
22. Patient has a known history of HIV infection (testing is not required);
23. Patient has any other concurrent sever and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial, or viral infections, etc.);
24. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks to starting study drug, or who have not fully recovered from side effects of such treatment
25. The following uses of corticosteroids are permitted: single doses, topical applications (e.g.: for rash), inhaled sprays (e.g.: for obstructive airways diseases), eye drops or local injections (e.g.: intra-articular);
26. Patient is currently receiving warfarin or other Coumadin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed;
27. Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer;
28. Patient who has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (exceptions include alopecia) and/or in whom ≥ 30-25% of the bone marrow was irradiated;
29. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery);
30. Patient has not recovered from all toxicities related to prior anticancer therapies to NCI-CTCAE version 4.03 Grade <1 (Exception to this criterion: patients with any grade of alopecia are allowed to enter the study);
31. Patient has a known hypersensitivity to any of the excipients of LEE011;
32. Prior ablative, radiation, resection, or transplant therapies less than 4 weeks before study registration;
33. Active gastrointestinal bleeding;
34. Allergy to iodine or gadolinium contrast that cannot be safely controlled with premedication;
35. Concurrent malignancy or malignancy within 3 years of study entry, with the exception of adequately treated basal or squamous cell carcinoma, non-melanomatous skin cancer or treated cervical cancer;
36. Contraindication to angiography or chemoembolization medications;
37. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after contraception and until the termination of gestation, confirmed by a positive hCG (Human chorionic gonadotropin) laboratory test;
38. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation. Highly effected contraception methods include:
39. Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
40. Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
41. Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient.
42. Combination of any of the two following (a+b or a+c or b+c) 43A-Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception; 45 B-Placement of an intrauterine device (IUD) or intrauterine system (IUS); 45 C-Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository in case of use of oral contraception, women should have been stable on the same pill before taking study treatment.

Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction. Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.

46-Sexually active males, unless they use a condom during intercourse while taking the drug, and for 21 days after stopping treatment of LEE011 -- should not father a child in this period. A condom is required to be used also by vasectomized male in order to prevent delivery of the drug via seminal fluid.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2020-09 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Beg, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- UT Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | LEE001 With Chemoembolization
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | LEE001 With Chemoembolization
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Non-Hispanic | 3
  Black or African American | 1
  Hispanic or Latino | 1
  Asian | 0
  Other | 0

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival
Description: CT Chest scans must be performed at baseline. CT-Chest/abdomen/pelvis must be performed every 8 weeks during the treatment phase (12 months). Once the patient has been discontinued from the study and enters the efficacy phase, radiological assessment (CT or MRI) will continue every 8 weeks until progression or for the first 12 months, whichever comes first. After a year, radiological (CT or MRI) assessments will be performed every 12 weeks for up to 1 year.
Time Frame: Every 8 weeks for up to 3 years.
Population: Data were not collected for this outcome due to early study termination
Arm/Group | LEE001 With Chemoembolization
Number analyzed (Participants) | 0

2. Secondary Outcome: Overall Survival
Description: CT Chest scans must be performed at baseline. CT-Chest/abdomen/pelvis must be performed every 8 weeks during the treatment phase (12 months). Once the patient has been discontinued from the study and enters the efficacy phase, radiological assessment (CT or MRI) will continue every 8 weeks until progression or for 3 years, whichever comes first. After a year, radiological (CT or MRI) assessments will be performed every 12 weeks for up to 3year.
Time Frame: Every 12 weeks for up to 3 years.
Population: Data were not collected for this outcome due to early study termination
Arm/Group | LEE001 With Chemoembolization
Number analyzed (Participants) | 0

3. Secondary Outcome: Number of Participants With Adverse Events
Description: Adverse events will be determined according to Common Terminology Criteria for Adverse Events (CTCAE) Version 4.0.
Time Frame: Each visit for up to 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | LEE001 With Chemoembolization
Number analyzed (Participants) | 5
Participants | 1

4. Secondary Outcome: Tolerability, as Measured by Number of Adverse Events
Description: The tolerability of LEE in combination with chemoembolization will be measured by number of adverse events.
Time Frame: At each patient visit while on LEE001 for up to 3 years
Measure: Number; unit: Adverse Events
Arm/Group | LEE001 With Chemoembolization
Number analyzed (Participants) | 5
Adverse Events | 1

5. Secondary Outcome: Objective Response Rate (ORR) Based on mRECIST and RECIST 1.1
Description: ORR was defined as number of participants with confirmed complete response (CR) or confirmed partial response (PR) according to the RECIST 1.1.
Time Frame: Every 8 weeks for 3 years
Measure: Count of Participants; unit: Participants
Arm/Group | LEE001 With Chemoembolization
Number analyzed (Participants) | 5
Participants | 2

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | LEE001 With Chemoembolization
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 1/5
Other Adverse Events (participants affected / at risk) | 0/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | LEE001 With Chemoembolization (N=5)
Hepatic infection (Infections and infestations) | 1 (1)

LIMITATIONS AND CAVEATS:
Data were not collected for some outcome due to early study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-19): https://cdn.clinicaltrials.gov/large-docs/19/NCT02524119/Prot_SAP_000.pdf